CLINICAL TRIAL: NCT01449552
Title: Temporary Clamping of Drains Combined With Tranexamic Acid Reduce Blood Loss After Total Knee Arthroplasty: A Prospective Randomized Controlled Trial.
Brief Title: Temporary Clamping of Drains Combined With Tranexamic Acid Reduce Blood Loss After TKA: A Prospective RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Keerati Charoencholvanich, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Si463/2007
Record Dates: First submitted 2011-10-05; First posted 2011-10-10 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): No clamp and placebo
  Interventions: Other: No clamp and placebo
- Group B (Experimental): Tranexamic acid
  Interventions: Drug: Tranexamic acid
- Group C (Experimental): Drain clamping
  Interventions: Procedure: Drain clamping
- Group D (Experimental): Drain clamping and tranexamic acid
  Interventions: Other: Drain clamping and tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — the drain was not clamped and the patient received tranexamic acid 10mg/kg intravenous 10 minutes before inflating the tourniquet and 10mg/kg intravenous three hours post-operative, and then tranexamic acid 250mg/capsule 2X3 orally for five days.
  Arms: Group B
Procedure: Drain clamping — the drain was clamped for three hours, released for three hours, then clamped for another three hours, and then released free for 48 hours. The patient received placebo (saline 10 minutes before surgery and three hours post-operative, and then an oral form of placebo 2X3 capsules for five days).
  Arms: Group C
Other: Drain clamping and tranexamic acid — the drain was clamped for three hours, released for three hours, then clamped for another three hours, and then released free for 48 hours. the patient received tranexamic acid 10mg/kg intravenous 10 minutes before inflating the tourniquet and 10mg/kg intravenous three hours post-operative, and then tranexamic acid 250mg/capsule 2X3 orally for five days.
  Arms: Group D
Other: No clamp and placebo — The drain was not clamped. The patient received placebo (saline 10 minutes before surgery and three hours post-operative, and then an oral form of placebo 2X3 capsules for five days).
  Arms: Group A

SUMMARY:
Total knee arthroplasty (TKA) may be associated with significant blood loss, and transfusion carries substantial risk of immunologic reaction and disease transmission. Several methods reportedly reduce postoperative blood loss and avoid homologous blood transfusion with traditional TKA approaches. Drain clamping was one of the widely used method and tranexamic acid administration was the recently adjuvant method to reduce blood loss in TKA. However, there were several regimens in either drain clamping or tranexamic acid administration reported in previous studies. Our objective was to compare the efficacy of our drain clamping protocol and/or tranexamic acid regimen for reducing blood loss and transfusion in TKA.

ELIGIBILITY:
Inclusion Criteria:

* The patients younger than 85 years with knee osteoarthritis

Exclusion Criteria:

* The patient diagnosed secondary osteoarthritis (eg, rheumatoid arthritis, posttraumatic arthritis, gouty arthritis, postseptic arthritis)
* High-risk medical comorbid patient
* The patient who was planed for simultaneous bilateral TKAs
* The patient who had history of thromboembolic disease or bleeding disorder
* The patient who was receiving anticoagulant drug treatment
* The patient who had allergy to tranexamic acid

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-06; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Postoperative blood loss | 48 hours after operation

SECONDARY OUTCOMES:
Number of blood transfusion | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Keerati Charoencholvanich, MD, Principal Investigator — Mahidol University

REFERENCES:
- [Derived] Chareancholvanich K, Siriwattanasakul P, Narkbunnam R, Pornrattanamaneewong C. Temporary clamping of drain combined with tranexamic acid reduce blood loss after total knee arthroplasty: a prospective randomized controlled trial. BMC Musculoskelet Disord. 2012 Jul 20;13:124. doi: 10.1186/1471-2474-13-124. PMID 22817651